CLINICAL TRIAL: NCT00585468
Title: Pharmacokinetic Profile of Myfortic (Enteric Coated Mycophenolate Sodium) in a Rapid Steroid Withdrawal Protocol in Combination With Tacrolimus in Stable Renal Transplant Recipients in the Fed and Fasting State
Brief Title: Pharmacokinetic Profile of Myfortic in Combination With Tacrolimus in Fed Versus Fasting State
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 15121; Award# CERL080AUS33 (Other Grant/Funding Number: Novartis Pharmaceuticals)
Record Dates: First submitted 2007-12-21; First posted 2008-01-03 (Estimated); Results first posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-04

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Myfortic - Fed State (Experimental): Mycophenolate sodium taken with a meal.
  Interventions: Drug: Myfortic
- Myfortic - Fasting State (Experimental): Mycophenolate sodium taken separately from food by 2 hours.
  Interventions: Drug: Myfortic

INTERVENTIONS:
Drug: Myfortic — Myfortic 720 mg orally twice daily
  Other Names: mycophenolate sodium; mycophenolic acid

SUMMARY:
Literature regarding the effect of food on the pharmacokinetic (PK) profile of enteric-coated mycophenolate sodium combined with tacrolimus and corticosteroid withdrawal is lacking. The objective of this study is to identify pharmacokinetic variables of mycophenolate sodium (Myfortic®) in the fed and fasting state in stable renal transplant patients on tacrolimus in combination with a rapid steroid withdrawal protocol.

DETAILED DESCRIPTION:
Mycophenolate sodium (Myfortic®) is an antiproliferative immunosuppressant used in renal transplantation. Mycophenolate sodium is formulated as an enteric coated tablet that releases mycophenolic acid (MPA) which in turn inhibits inosine monophosphate dehydrogenase (IMPDH). Through inhibition of IMPDH, the de novo pathway of purine synthesis, which T and B lymphocytes rely on for proliferation, is blocked. The pharmacokinetic profile of mycophenolate sodium has mainly been studied in combination with cyclosporine and steroids. There is little information on the pharmacokinetics of mycophenolate sodium in combination with tacrolimus and currently no published information in steroid withdrawal. All current published data on the pharmacokinetics of MPA have been in patients receiving chronic corticosteroids as part of their immunosuppression regimen. As immunosuppression minimization, and especially corticosteroid withdrawal, become more popular it is important to understand how mycophenolate sodium and its metabolites behave in a two-drug maintenance immunosuppression regimen. The study will assess the pharmacokinetic profile of mycophenolate sodium in patients on tacrolimus dose adjusted based on levels, and a steroid withdrawal protocol.

Renal transplant patients will act as their own controls in a randomized crossover design with pharmacokinetic profiles occurring at two different time points. Immunosuppression will consist of induction therapy with maintenance immunosuppression consisting of tacrolimus plus mycophenolate sodium. Corticosteroids will be withdrawn per institutional protocol within the first week post transplant.

Approximately 3-4 weeks post transplant, patients that met enrollment criteria and have consented to participate in the study will be instructed to take 720 milligrams of mycophenolate sodium orally twice daily for one week either separated from food by two hours (fasting state) or with a meal (fed state). After one week, patients will be admitted for approximately 24 hours where they will continue to receive mycophenolate sodium with or without food. During this period, blood samples will be drawn at 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12 hours following the dose to evaluate levels of mycophenolic acid (MPA) and mycophenolic acid glucuronide (MPAG). After 24 hours, patients will be discharged with instructions to take mycophenolate sodium in the opposite manner (fed or fasting state) than they had the week before. At the end of the second week the patients will return for a second PK evaluation with blood collection at the same time points following mycophenolate sodium dosing.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant recipients greater than 18 years of age, who have given written consent

Exclusion Criteria:

* Taking medications that may alter the metabolism of tacrolimus or mycophenolate sodium
* Experienced an acute rejection episode prior to the pharmacokinetic profile collection
* Serum creatinine >2 mg/dL
* Neutropenia (Absolute Neutrophil Count < 1.3x10^3/mL)
* Received a previous transplant other than a kidney
* Receiving chronic steroids at time of transplant
* Known hypersensitivity to tacrolimus, mycophenolate mofetil, mycophenolate sodium, mycophenolic acid or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fuad Shihab, MD, Principal Investigator — University of Utah
Locations (1):
- Univ of Utah-Solid Organ Transplant, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Arns W, Breuer S, Choudhury S, Taccard G, Lee J, Binder V, Roettele J, Schmouder R. Enteric-coated mycophenolate sodium delivers bioequivalent MPA exposure compared with mycophenolate mofetil. Clin Transplant. 2005 Apr;19(2):199-206. doi: 10.1111/j.1399-0012.2004.00318.x. PMID 15740555
- [Background] Kaplan B, Meier-Kriesche HU, Minnick P, Bastien MC, Sechaud R, Yeh CM, Balez S, Picard F, Schmouder R. Randomized calcineurin inhibitor cross over study to measure the pharmacokinetics of co-administered enteric-coated mycophenolate sodium. Clin Transplant. 2005 Aug;19(4):551-8. doi: 10.1111/j.1399-0012.2005.00387.x. PMID 16008604
- [Background] Zucker K, Rosen A, Tsaroucha A, de Faria L, Roth D, Ciancio G, Esquenazi V, Burke G, Tzakis A, Miller J. Unexpected augmentation of mycophenolic acid pharmacokinetics in renal transplant patients receiving tacrolimus and mycophenolate mofetil in combination therapy, and analogous in vitro findings. Transpl Immunol. 1997 Sep;5(3):225-32. doi: 10.1016/s0966-3274(97)80042-1. PMID 9402690
- [Background] van Gelder T, Klupp J, Barten MJ, Christians U, Morris RE. Comparison of the effects of tacrolimus and cyclosporine on the pharmacokinetics of mycophenolic acid. Ther Drug Monit. 2001 Apr;23(2):119-28. doi: 10.1097/00007691-200104000-00005. PMID 11294511

RESULTS

PARTICIPANT FLOW:
Groups:
- Fed State First, Then Fasting State: 720 milligrams (mg) mycophenolate sodium orally twice daily with a meal for one week in the first intervention period, followed by one week of 720 mg mycophenolate sodium orally twice daily separated by food by 2 hours in the second intervention period.
- Fasting State First, Then Fed State: 720 mg mycophenolate sodium orally twice daily separated from food by 2 hours for one week in the first intervention period, followed by one week of 720 mg mycophenolate sodium orally twice daily with a meal in the second intervention period.
Period: First Intervention
Arm/Group | Fed State First, Then Fasting State | Fasting State First, Then Fed State
Started | 10 | 11
Completed | 9 | 10
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Second Intervention
Arm/Group | Fed State First, Then Fasting State | Fasting State First, Then Fed State
Started | 9 | 10
Completed | 9 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to the Fed State first and to the Fasted State first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 21
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 21

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Mycophenolic Acid (MPA)
Time Frame: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Myfortic - Fed State | Myfortic - Fasting State
Number analyzed (Participants) | 19 | 19
micrograms per milliliter | 12.8 (6.7) | 18.7 (7.7)
Statistical Analysis 1: Comparison: Myfortic - Fed State vs Myfortic - Fasting State; Test type: Superiority or Other; p = 0.0163, t-test, 2 sided

2. Primary Outcome: Minimum Observed Plasma Concentration (Cmin) of Mycophenolic Acid (MPA)
Time Frame: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Myfortic - Fed State | Myfortic - Fasting State
Number analyzed (Participants) | 19 | 19
micrograms per milliliter | 2.2 (0.6) | 1.7 (0.8)
Statistical Analysis 1: Comparison: Myfortic - Fed State vs Myfortic - Fasting State; Test type: Superiority or Other; p = 0.039, t-test, 2 sided

3. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Mycophenolic Acid (MPA)
Time Frame: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Measure: Median (Full Range); unit: hours
Arm/Group | Myfortic - Fed State | Myfortic - Fasting State
Number analyzed (Participants) | 19 | 19
hours | 5 [0 to 10] | 3 [0 to 8]

4. Primary Outcome: Area Under the Curve (AUC) From Time Zero to 12 Hours Post-Dose [AUC (0-12)] of Mycophenolic Acid (MPA)
Description: AUC (0-12) = Area under the plasma concentration versus time curve from time zero (pre-dose) to 12 hours post-dose, measured in microgram-hours per milliliter (mcg*h/mL)
Time Frame: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Myfortic - Fed State | Myfortic - Fasting State
Number analyzed (Participants) | 19 | 19
mcg*h/mL | 56.5 (15.2) | 63.9 (15.5)
Statistical Analysis 1: Comparison: Myfortic - Fed State vs Myfortic - Fasting State; Test type: Superiority or Other; p = 0.146, t-test, 2 sided

5. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Mycophenolic Acid Glucuronide (MPAG)
Time Frame: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Myfortic - Fed State | Myfortic - Fasting State
Number analyzed (Participants) | 19 | 19
micrograms per milliliter | 104.9 (35.7) | 113.0 (36.5)
Statistical Analysis 1: Comparison: Myfortic - Fed State vs Myfortic - Fasting State; Test type: Superiority or Other; p = 0.4937, t-test, 2 sided

6. Primary Outcome: Minimum Observed Plasma Concentration (Cmin) of Mycophenolic Acid Glucuronide (MPAG)
Time Frame: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Measure: Mean (Standard Deviation); unit: micrograms per milliliter
Arm/Group | Myfortic - Fed State | Myfortic - Fasting State
Number analyzed (Participants) | 19 | 19
micrograms per milliliter | 59.4 (24.9) | 57.0 (23.0)
Statistical Analysis 1: Comparison: Myfortic - Fed State vs Myfortic - Fasting State; Test type: Superiority or Other; p = 0.9669, t-test, 2 sided

7. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Mycophenolic Acid Glucuronide (MPAG)
Time Frame: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Measure: Median (Full Range); unit: hours
Arm/Group | Myfortic - Fed State | Myfortic - Fasting State
Number analyzed (Participants) | 19 | 19
hours | 3 [0 to 11] | 3 [1 to 7]

8. Primary Outcome: Area Under the Curve From Time Zero to 12 Hours Post-Dose [AUC (0-12)] of Mycophenolic Acid Glucuronide (MPAG)
Description: as for outcome 4
Time Frame: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 hours post-dose
Measure: Mean (Standard Deviation); unit: mcg*h/mL
Arm/Group | Myfortic - Fed State | Myfortic - Fasting State
Number analyzed (Participants) | 19 | 19
mcg*h/mL | 967.5 (364.0) | 962.2 (289.6)
Statistical Analysis 1: Comparison: Myfortic - Fed State vs Myfortic - Fasting State; Test type: Superiority or Other; p = 0.9607, t-test, 2 sided

ADVERSE EVENTS:
Description: Adverse events were not collected in this study
Arm/Group | Myfortic - Fed State | Myfortic - Fasting State
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes